CLINICAL TRIAL: NCT00407875
Title: A Randomized Phase II Study Comparing Intensity Modulated External Beam Radiation Therapy (IMRT) Versus Permanent Interstitial Prostate Brachytherapy (PIPB) for Low Risk and Low-tier Intermediate Risk Prostate Cancer
Brief Title: Intensity Modulated Versus Interstitial - Radiation Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Principal Investigator, James Morris, Radiation Oncologist, British Columbia Cancer Agency
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMVI-RT
Record Dates: First submitted 2006-12-01; First posted 2006-12-05 (Estimated); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: Prostate Cancer
Keywords: Prostate; Cancer; Radiation
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms

ARMS (2):
- Permanent interstitial prostate brachytherapy (PIPB) (Active Comparator): patient will undergo permanent interstitial prostate brachytherapy (PIPB) using a transperineal approach to deliver 125Iodine Rapidstrand® seeds at the facilities of the British Columbia Cancer Agency (BCCA) by one or more of the certified prostate brachytherapists in the BCCA Prostate Brachytherapy Program. The minimum peripheral dose (MPD) to the prostate gland of the implant will be 144 Gy as per TG 43 protocol. A modified peripheral loading technique will be utilized in an effort to maintain the periurethral dose to < 150% of the MPD. Within 48 hours of the implant, the patient will undergo a day 0 CT scan of the pelvis to assess post implant dosimetry using the standard BCCA protocol.
  Interventions: Procedure: Intensity Modulated External Beam Radiation Therapy
- Intensity modulated external beam radiation therapy (IMRT) (Experimental): patient will undergo a course of intensity modulated external beam radiation therapy (IMRT) to a volume encompassing the prostate gland. The total radiation dose will be 70 Gy delivered in 28 fractions, so that the minimum dose to the PTV is 70 Gy, with CT simulation used for planning the treatment. Prior to starting the course of IMRT, fiducial markers will be placed in the prostate to assist in localization of the prostate for planning and quality assurance during treatment.
  Interventions: Procedure: Intensity Modulated External Beam Radiation Therapy

INTERVENTIONS:
Procedure: Intensity Modulated External Beam Radiation Therapy

SUMMARY:
Purpose:

The purpose of this trial is to compare two different treatment options for patients with low risk and low-tier intermediate risk prostate cancer. The two treatment arms being compared in this study are: (control arm) permanent interstitial prostate brachytherapy (PIPB) VERSUS (experimental arm) intensity modulated external beam radiation therapy (IMRT).

Hypothesis:

The acute and late toxicities experienced by patients in the experimental arm (IMRT) are not significantly worse then the toxicities experienced by patients in the control arm (PIPB).

DETAILED DESCRIPTION:
Justification:

Patients with low risk and low-tier intermediate risk prostate cancer have a number of different standard treatment options to chose from that include a radical prostatectomy, conventional external beam radiotherapy (EBRT), or permanent interstitial prostate brachytherapy (PIPB). Each of these treatment options have good outcomes, although they are known to have a small risk of complications associated with each of them. Unfortunately, these treatment options have never been directly compared and therefore it is difficult to determine how these treatment options compare with respect to overall outcomes and toxicity.

A recent analysis from the BC Cancer Agency suggested that patients treated with conventional EBRT within the Agency had inferior outcomes compared to PIPB. This data, as well as other indirect evidence, suggest that conventional EBRT may be a suboptimal treatment option compared to PIPB. Intensity modulated external beam radiotherapy (IMRT) is a new technology that allows for the delivery of high doses of radiation that tightly conforms to the target and limits the dose to surrounding critical structures. Although IMRT is currently a standard therapeutic option that is utilized in other cancer sites at the BC Cancer Agency, it has not been utilized in prostate cancer yet. Recent evidence has confirmed that this experimental therapy is able to allow for the safe escalation of dose for prostate cancer patients, which may lead to improved outcomes, without increasing toxicity. There is no current evidence that side effects and complication risks associated with IMRT are associated with any serious risk of increased toxicity, although this continues to be studied.

This study will compare this new therapeutic approach (IMRT) directly with a standard treatment option for prostate cancer patients (PIPB). This trial will allow us to determine how the toxicities of these treatments compare with each other and, if successful, will potentially lead to a larger study which will analyse how the outcomes of these therapeutic interventions compare. We hope that this trial will make an important contribution to the care and future management of patients with prostate cancer.

Objectives:

Primary Objective:

The primary end point of this study is the acute and late toxicities of the therapeutic interventions.

Secondary Objectives:

This trial is also intended to determine:

* The willingness of eligible patients to be randomized to the treatment interventions.
* Obstacles to accrual that need to be addressed.
* Testing our ability to meet accrual targets.
* Checking quality assurance benchmarks for IMRT and PIPB procedures.
* Discovering and relieving bottlenecks in IMRT planning and procedures.
* Quality of life.
* Pathological local control.
* Biochemical relapse-free survival.
* Metastasis-free survival.
* Overall survival.

Research Method:

The patients will be randomly assigned with equal probability to one of two treatment arms:

Arm 1 (Control Arm) - Permanent interstitial prostate brachytherapy (PIPB). Arm 2 (Experimental Arm) - Intensity modulated external beam radiation therapy (IMRT).

Statistical Analysis:

Primary Endpoints:

Acute GI grade 3 or higher toxicity. Acute GU grade 3 or higher toxicity. Late GI grade 3 or higher toxicity. Late GU grade 3 or higher toxicity.

Secondary Endpoints:

All acute and late toxicities. Quality of life scores (Using the expanded prostate cancer index composite - EPIC).

Pathological local control. Biochemical relapse-free survival (using Phoenix definition). Metastasis-free survival. Overall survival.

Planned sample size: 50 patients in total (i.e. 25 patients in each treatment arm).

Statistical analysis:

The two groups will be compared with respect to their primary and secondary endpoints. Appropriate statistical analysis using a student t test for a statistical difference in crude rates of grade 3 or higher toxicity between the two treatment arms will be performed. All endpoints will be analysed for crude event rates with 95% confidence intervals for each group.

With a sample size of only 50 patients, this trial is not powered to detect differences in the incidence of common self-limited side effects and adverse reactions compared to standard therapy. For this reason, the trial's limited power is augmented by a Trial Safety Committee (TSC) which is bound by rules that require suspension/ termination of trial accrual in the event of major complications (See Section 8.3 of Data Monitoring - Human Ethics Application for Clinical Study or Part I: Section 5.3 on page 11 of the protocol).

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically proven adenocarcinoma of the prostate.
2. Registration must occur within 20 weeks of biopsy.
3. History and physical examination within 8 weeks prior to randomization.
4. Patients must have either low risk or low-tier intermediate risk prostate cancer (Low risk must have all of: clinical stage <= T2b, Gleason score <= 6, and initial PSA <= 10; Low-tier intermediate risk must have: clinical stage <= T2c, < 50% positive biopsy cores, AND EITHER Gleason score = 7 and initial PSA <= 10 OR Gleason score <= 6 and initial PSA > 10 and <= 15.)
5. Patients must have a ECG, PSA, TTT, CBC, electrolytes, Cr, INR, PTT, and random glucose within 2 weeks of registration.
6. Patients must be fit for general or spinal anesthetic.
7. Patients must have an estimated life expectancy of at least 10 years.
8. Patients must have an ECOG performance status of 0 - 2.
9. Patients must have no contraindications for high dose pelvic irradiation or transperineal interstitial brachytherapy.
10. Patients must not have received prior radiation therapy to the pelvis.
11. Patients must have no history of inflammatory bowel disease.
12. Patients must not have received prior hormonal therapy or chemotherapy.
13. Patients must not have any hormonal therapy planned as part of the therapeutic intervention.
14. Patients must have prostate volumes < 60 cm3 on transrectal ultrasound.
15. Patients must not have received prior surgical treatment for prostate cancer including TURP, TURB, cryotherapy, laser ablation or microwave therapy.
16. Patients on coumadin therapy must be able to stop therapy safely for at least 12 days.
17. Patients must have an International Prostate Symptom Score (IPSS) of less than 20.
18. Patients must have no history of previous malignancies, except non-melanoma skin tumors.
19. Patients must have a body mass index (BMI) of <= 32.

Exclusion Criteria:

Those patients who do not meet the inclusion criteria described above will be excluded from participation.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-03; Primary Completion 2008-03 (Actual); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
The primary end point of this study is the acute and late toxicities of the therapeutic interventions. | Through study completion. Approximately 5 years.

SECONDARY OUTCOMES:
The willingness of eligible patients to be randomized to the treatment interventions. | 1 year
Obstacles to accrual that need to be addressed. | 1 year
Testing our ability to meet accrual targets. | 1 year
Checking quality assurance benchmarks for IMRT and PIPB procedures. | 1 year
Quality of life based on urinary function, bowel habits, sexual function, and hormonal function | Assessed at 6 weeks, 6, 9, 12, 18, 24 ,30, 36 months. Then annually until end of participation
Pathological local control. | Assessed at 28 months
Biochemical relapse-free survival. | Assessed at every clinic visit and every 6 months
Metastasis-free survival. | Assessed at every clinic visit until end of participation. Approximately 10 years.
Overall survival. | Assessed at every clinic visit until end of participation. Approximately 10 years.

CONTACTS AND LOCATIONS:
Overall Officials: William J Morris, MD, Principal Investigator — British Columbia Cancer Agency
Locations (1):
- BC Cancer Agency, Vancouver, British Columbia, Canada